CLINICAL TRIAL: NCT05857241
Title: Therapeutic Fasting and Immune Aging: A Pilot Study of Tolerance
Brief Title: Therapeutic Fasting and Immune Aging
Acronym: JÛVENILE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21CH028; 2023-A00390-45 (Other: ANSM)
Record Dates: First submitted 2023-04-04; First posted 2023-05-12 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Fasting; Diet, Healthy
Keywords: Fasting mimicking diet; Aged; immunology; immunosenescence; tolerance
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fasting mimicking diet (FMD) (Experimental): patients aged 65 and over, institutionalized in Long Term Care Units (USLD) or Establishments for the elderly (EHPAD).
  Interventions: Dietary Supplement: Fasting mimicking diet (FMD)

INTERVENTIONS:
Dietary Supplement: Fasting mimicking diet (FMD) — D1 will correspond to a "pre-fasting" phase, with about 800 kcal of intake (approximately 40% of normal caloric intake) from a mono-nutrient diet (fruit, rice or potato according to the patient's preferences). Then D2 and D3 will correspond to the days of actual fasting, with 200-350 kcal of intake (10-18% of normal caloric intake) in the form of 100 ml of broth or vegetable juice (with a teaspoon of linseed oil) three times a day, and vaccination will take place on D4, after returning to a normal diet. 2 to 3 liter of water or unsweetened drink per day is required.Laxatives (unsweetened) will be prescribed and can be taken as during the fasting period.

SUMMARY:
Immunosenescence is the age-related decline of the immune system, involving a state of chronic inflammation and a decrease in the diversity/adaptability of the lymphocyte repertoire. The consequences of immunosenescence are multiple, including increased susceptibility to infections and poorer vaccine responses.

DETAILED DESCRIPTION:
In order to fight against immunosenescence, many therapeutics are envisaged, with the aim of restoring, renewing and/or reprogramming the immune system. Among these leads, therapeutic fasting, and in particular the "fasting mimicking diet" (FMD), seems to modify the reprogramming and renewal of the immune system with, on the one hand, the elimination of inefficient "overactivated" cells and, on the other hand, the activation of hematopoietic stem cells. FMD consists of a significant reduction in food intake, limited to 3-5 days/month. The FMD seems to be the best compromise between efficacy and tolerance (already evaluated in humans, including oncology).

ELIGIBILITY:
Inclusion Criteria :

* Patient affiliated or entitled to a social security scheme
* Residing in a Long-Term Care Unit (LTCU) or a Facility for the Elderly Dependent (EHPAD)
* A person deemed a priori, by the geriatrician member of the monitoring committee, to be capable of following the dietary recommendations required for the study.
* A person deemed a priori, by the clinician in charge, to be able to follow the dietary recommendations required by the study.
* Patient who has received informed information about the study and has co-signed a consent to participate in the study with the investigator.

Exclusion Criteria :

* Inability and/or unwillingness to follow dietary recommendations and/or perform follow-up examinations required for the study
* Iso-resource group 1 or 2 according to the AGGIR grid
* BMI < 18.5 kg/m2 or recent weight loss > 5% in 1 month or recent weight loss > 10% in 6 months from previous weight
* Albuminemia < 30g/l
* All swallowing disorders requiring a specific diet.
* Influenza vaccination received prior to inclusion
* Episode of influenza or suspected influenza during the 2020-2021 season and prior to inclusion
* Any acute medical or surgical event less than 2 weeks prior to inclusion
* Presence of systemic inflammatory or autoimmune disease
* Presence of an innate or acquired immune deficiency (including taking immunosuppressive treatment)
* Presence of a chronic disease which, according to the physician, makes the follow-up of a "fasting diet" and/or the consumption of large amounts of liquids (cf. fasting diet modalities) risky (e.g. insulin-dependent or insulin-requiring diabetes, severe heart failure, severe kidney failure, active cancer, significant undernutrition...) or impossible (e.g. advanced neurodegenerative pathology).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
rate of premature discontinuation of the fasting-mimicking diet | between Day 14 and Day 21
  measurement of the rate of occurrence of a clinical event considered to require discontinuation of the fasting diet :
  The occurrence of a clinical event considered to require discontinuation of the fasting diet will be defined as the presence between D14 and D21 of at least one of the following conditions:
  * Weight loss > 5%,
  * Hypoglycemia < 0.5 g/l (< 2.8 mmol/l),
  * Hypothermia < 35°C,
  * Heart rate < 50 beats per minute, checked twice at 15 minute intervals,
  * Low systolic blood pressure < 90 mmHg or > 200 mmHg; or diastolic blood pressure < 60 mmHg or > 110 mmHg; or mean blood pressure < 70 mmHg, checked twice at 15-minute intervals,
  * Increase of 5 points on the visual analog pain scale between D14 and D21,
  * A score of 1 on the EVIBE visual analog scale (instantaneous assessment of well-being) between D14 and D21,
  * Any serious acute clinical event (fall with serious traumatic consequence, acute medical or surgical condition).

SECONDARY OUTCOMES:
serious and non-serious adverse events reported | Between day 0 to day 42
  Comparison of the nature and frequency of serious and non-serious adverse events reported from D0 to D13 (pre fasting diet phase), D14 to D16 (fasting diet phase) and D17 to D42 (post fasting diet phase)
composite outcome: evolution of biological biochemic parameters | Day 0 to Day 42
  Evolution of measurements of blood glucose, ketones, albumin, prealbumin and IGF-1 Unit of measure : ng/ml
composite outcome: evolution of biological blood parameters | Day 0 to Day 42
  Evolution of the measurement of the blood total lymphocyte count (CD4, CD8, CD19, naive, effectors, memories, regulators, etc.).
  Unit of measure : %
composite outcome: evolution biological inflammatory parameters | Day 0 to Day 42
  Evolution of inflammatory markers (CRP, IL1, IL6, TNFalpha) Unit of measure : ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Baptiste GRAMONT, MD, Principal Investigator — Baptiste.Gramont@chu-st-etienne.fr
Locations (5):
- France (5):
  - EHPAD Claudinon, Le Chambon-Feugerolles
  - EHPAD Les Cèdres Malataverne, Malataverne
  - CHU de Saint-Etienne, Saint-Etienne
  - EHPAD de la Talaudière, la Rivière, la Croix de l'Horme, Saint-Etienne
  - EHPAD La M.R.L, Saint-Just-Saint-Rambert

IPD SHARING:
Plan to Share IPD: No